CLINICAL TRIAL: NCT05503797
Title: A Phase 2 Master Protocol to Assess the Efficacy and Safety of FORE8394, an Inhibitor of BRAF Class 1 and Class 2 Alterations, in Participants With Cancer Harboring BRAF Alterations
Brief Title: A Study to Assess the Efficacy and Safety of FORE8394 in Participants With Cancer Harboring BRAF Alterations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fore Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F8394-201; 2024-513578-23-00 (EU CTIS Number); 2022-000627-20 (EudraCT Number)
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Cancer Harboring BRAF Alterations; HGG; LGG; Solid Tumors
Keywords: BRAF alterations; BRAF Fusions; BRAF V600E; BRAF Class 1; BRAF Class 2; High grade glioma; low grade glioma; HGG; LGG; Solid tumors
MeSH Terms: conditions — Glioma | interventions — PLX8394

STUDY DESIGN:
Intervention Model Description: All four open-label single-arm subprotocols will enroll patients independently of one another, in parallel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Subprotocol A (Experimental): Participants with unresectable, locally advanced or metastatic solid tumors or primary CNS tumors harboring BRAF fusions will receive plixorafenib which will be increased as tolerated, continuously in 3-week cycles until disease progression, unacceptable toxicity, or other reason for withdrawal.
  Interventions: Drug: Plixorafenib
- Subprotocol B (Experimental): Participants with recurrent primary CNS tumors harboring BRAF V600E mutations will receive plixorafenib, continuously in 3-week cycles until disease progression, unacceptable toxicity, or other reason for withdrawal.
  Interventions: Drug: Plixorafenib
- Subprotocol C (Experimental): Participants with advanced, rare, non-CNS solid tumors harboring BRAF V600E mutations will receive plixorafenib, continuously in 3-week cycles until disease progression, unacceptable toxicity, or other reason for withdrawal.
  Interventions: Drug: Plixorafenib
- Subprotocol D (Experimental): Participants with BRAF V600E-mutated advanced solid tumors will receive plixorafenib until disease progression, unacceptable toxicity, or other reason for withdrawal.
  Interventions: Drug: Plixorafenib

INTERVENTIONS:
Drug: Plixorafenib — Oral tablets
  Other Names: FORE8394; PLX8394

SUMMARY:
The objective of this Master Protocol is to evaluate the efficacy and safety of plixorafenib in participants with locally advanced or metastatic solid tumors, or recurrent or progressive primary central nervous system (CNS) tumors harboring BRAF fusions, or in participants with rare BRAF V600-mutated solid tumors, melanoma, thyroid, or recurrent primary CNS tumors.

ELIGIBILITY:
Inclusion Criteria

Subprotocol A:

1. Male and female, ≥10 years of age, and weighing ≥30 kg.
2. Histologic diagnosis of a solid tumor or primary CNS tumor.
3. Documentation of BRAF gene fusion in tumor and/or blood detected by an analytically validated test by DNA sequencing or RNA (transcriptome) sequencing.
4. Have an archival tissue sample available meeting protocol requirements.
5. Consent to provide scan(s) prior to baseline to assess change in tumor trajectory.
6. Received all available standard therapy, is intolerant to available therapies, or the investigator has determined that treatment with standard therapy is not appropriate.
7. All adverse events related to prior therapies (chemotherapy; radiotherapy; surgery) must have resolved to Grade 1 or baseline.

Subprotocol B:

1. Male and female, ≥10 years of age, and weighing ≥30 kg.
2. Histological diagnosis of a primary CNS tumor, including but not limited to the following:

   1. Adults (≥18 years) with Grade 1-4 glioma or glioneuronal tumor (including glioblastoma, anaplastic astrocytoma, high grade astrocytoma with piloid features, pilocytic astrocytoma, gliosarcoma, anaplastic pleomorphic xanthoastrocytoma, anaplastic oligodendroglioma, anaplastic oligoastrocytoma, not otherwise specified [NOS], ganglioglioma, or recurrent LGG). OR
   2. Pediatric patients (10-17 years of age) with a Grade 3 or 4 glioma or glioneuronal tumor, including those with a prior, histologically confirmed, diagnosis of a low-grade glioma or glioneuronal tumor and now have radiographic or histopathological findings consistent with WHO [2021] Grade 3 or 4 primary CNS tumor.
   3. Participants must have unresectable, locally advanced or metastatic disease that:

   i. Had prior treatment with radiotherapy and/or first-line chemotherapy or concurrent chemoradiation therapy OR
   * Note: Participants who have a WHO Grade 3 or 4 glioma for whom chemotherapy and/or radiotherapy is not considered standard of care may remain eligible for the study.

   ii. Is intolerant to available therapies OR iii. The investigator has determined that treatment with standard therapy is not appropriate.
3. Documented BRAF V600E mutation in tumor and/or liquid biopsy detected by an analytically validated test at CLIA or CLIA-equivalent laboratory approved by sponsor or sponsor-designated central test.
4. An archival tissue sample available meeting protocol requirements, or fresh biopsy is required if the archival sample is not available for retrospective confirmation test.
5. Consent to provide scan(s) prior to baseline to assess change in tumor trajectory.
6. Measurable disease based upon specified response criteria, as determined by the radiographic BICR.
7. All adverse events related to prior therapies (eg, chemotherapy, radiotherapy, surgery) must have resolved to Grade 1 or baseline.
8. Participants who are receiving corticosteroid treatment must be on a stable or decreasing dose of ≤8 mg/day of dexamethasone or equivalent corticosteroid treatment for 7 days prior to first dose of study treatments.

Subprotocol C:

1. Male and female, ≥10 years of age, and weighing ≥30 kg.
2. Histologic diagnosis of a rare BRAF V600E-mutated solid tumor that is unresectable, locally advanced or metastatic.
3. Measurable disease on CT, MRI, or physical exam
4. Documented BRAF V600E mutation in tumor and/or liquid biopsy detected by an analytically validated test.
5. Have an archival tissue sample available meeting protocol requirements.
6. Consent to provide scan(s) prior to baseline to assess change in tumor trajectory
7. Received all available standard therapy, is intolerant to available therapies, or the investigator has determined that treatment with standard therapy is not appropriate.

Subprotocol D:

1. Male and female, 18 - 65 years of age.
2. Histologic diagnosis of a solid tumor harboring a BRAF V600E mutation and not eligible for other subprotocols.
3. Measurable disease on CT, MRI, or physical exam.
4. Evidence of BRAF V600E mutation in tumor and/or blood detected by genomic tests.
5. Consent to provide a tumor biopsy.
6. Willingness to comply with the ECG substudy procedures.
7. All adverse events related to prior therapies (chemotherapy; radiotherapy; surgery) must have resolved to Grade 1 or baseline.

Exclusion Criteria:

Subprotocol A:

1. Prior treatment with RAF/BRAF inhibitors active for Class 2 BRAF alterations for advanced unresectable or metastatic disease.
2. Prior treatment with a MEK inhibitor.
3. Tyrosine kinase inhibitor(s) and/or targeted therapies are allowed (other than BRAF/MAPK pathway inhibitors per Exclusion Criteria 3 and 4) and will be restricted to no more than the number of lines of therapy that are consistent with standard treatment guidelines.
4. Malignancy with co-occurring activating RAS mutation(s) at any time.
5. Uncontrolled intercurrent illness that would limit compliance with study requirements.
6. HIV infection with exceptions; discuss with treating physician.
7. Have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral plixorafenib or cobicistat (such as ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, and small bowel resection).
8. Grade ≥2 changes in AST, ALT, GGT, or bilirubin attributed to prior immune checkpoint inhibitor treatment are exclusionary, even if resolved.

Subprotocol B:

1. Prior treatment with BRAF, ERK, and/or MEK inhibitor(s).
2. Known or suspected neurofibromatosis-1 (NF-1) and/or RAS related gene alterations.
3. Uncontrolled intercurrent illness that would limit compliance with study requirements.
4. Active infection requiring systemic therapy.
5. HIV infection with exceptions; discuss with treating physician.
6. Have impairment of GI function or GI disease that may significantly alter the absorption of oral plixorafenib (such as ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
7. Grade ≥ 2 changes in AST, ALT, gamma-glutamyl transaminase (GGT), or bilirubin attributed to prior immune checkpoint inhibitor treatment are exclusionary, even if resolved.

Subprotocol C:

1. Diagnosis of colorectal adenocarcinoma or pancreatic ductal adenocarcinoma (neuroendocrine or acinar tumors are eligible).
2. Diagnosis of BRAF V600E-mutated cutaneous melanoma, papillary thyroid cancer, or NSCLC.
3. Participant has CNS metastases.
4. Prior treatment with BRAF, ERK, and/or MEK inhibitor(s), unless otherwise specified for specific tumor types (i.e. low grade serous or borderline ovarian cancer).
5. Known or suspected neurofibromatosis-1 (NF-1) and/or RAS related gene alterations.
6. Participants with prostate, breast, or gynecologic cancers with known activating mutations that lead to constitutive hormone receptor activation (AR-V7, ESR1).
7. Uncontrolled intercurrent illness that would limit compliance with study requirements.
8. Active infection requiring systemic therapy.
9. HIV infection with exceptions; discuss with treating physician.

Subprotocol D:

1. Known or suspected neurofibromatosis-1 (NF-1) and/or RAS related gene alterations or other co-occurring driver mutations.
2. Participant has a non-CNS solid tumor with CNS metastases.
3. Uncontrolled intercurrent illness that would limit compliance with study requirements.
4. Active infection requiring systemic therapy.
5. HIV infection with exceptions; discuss with treating physician.
6. Use or anticipate the need for medications with known risk for QT-prolonging potential and Torsades de Pointes.
7. History of acute or chronic cardiovascular disease or surgery, hypertension, with systolic blood pressure >160mm HG, history of QTc abnormalities, or clinical significantly ECG abnormalities.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) (Subprotocols A, B and C) | Up to approximately 4 years
  ORR will be determined by standard tumor response criteria by blinded independent central review (BICR).
Pharmacokinetics (Subprotocol D) | Up to approximately 4 years
  Systemic exposure of plixorafenib measured by Cmax and AUC

SECONDARY OUTCOMES:
Duration of Response (DOR) by BICR (Subprotocols A, B and C) | Up to approximately 4 years
  DOR will be determined by standard tumor response criteria per BICR (subprotocols A-C)
ORR per Investigator Assessment | Up to approximately 4 years
  ORR will be determined by standard tumor response criteria by Investigator Assessment.
DOR per Investigator Assessment | Up to approximately 4 years
  DOR will be determined by standard tumor response criteria.
Percentage of Participants with DOR at 6 months, 12 months, and 18 months | 6 months, 12 months and 18 months
Time to Response by BICR (Subprotocols A, B and C) | Up to approximately 4 years
Progression Free Survival (PFS) by BICR (Subprotocols A, B and C) | Up to approximately 4 years
PFS per Investigator's Assessment | Up to approximately 4 years
Overall Survival | Up to approximately 4 years
Percentage of Participants with PFS at 6 months, 12 months and 24 months | 6 months, 12 months and 24 months
  BICR (Subprotocols A, B and C) and by Investigator Assessment (Subprotocols A, B, C and D)
Disease Control Rate (DCR) | Up to approximately 4 years
Number of Participants who Experience Treatment-emergent Adverse Events (TEAEs) | Up to approximately 4 years
Plasma Concentrations of Plixorafenib | Up to approximately 4 years
Plasma Concentrations of Plixorafenib Metabolites | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Locations (64):
- United States (26):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of California Los Angeles Rheumatology, Westwood, Los Angeles, California
  - Norwalk Hospital, Norwalk, Connecticut
  - University of Miami Hospital and Clinics, Miami, Florida
  - The John Hopkins Hospital, Baltimore, Maryland
  - Maryland Oncology Hematology- Columbia, Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - St. Luke's Hospital, Duluth, Minnesota
  - Mosaic Life Care at Saint Joseph - Medical Center, Saint Joseph, Missouri
  - Nebraska Cancer Specialists - Midwest Cancer Center - Legacy, Omaha, Nebraska
  - Overlook Medical Center, Summit, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Atrium Health Wake Forest Baptist - Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Taylor Cancer Research Center, Maumee, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Lifespan Cancer Institute - Rhode Island Hospital, Providence, Rhode Island
  - SCRI - TriStar Medical Group Children's Specialists, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Baylor Scott & White Medical Center, Temple, Texas
  - University of Washington School of Medicine, Seattle, Washington
  - West Virginia University Health Sciences Campus, Morgantown, West Virginia
- Australia (4):
  - Newcastle Private Hospital, New Lambton Heights, New South Wales
  - Orange Health Service, Orange, New South Wales
  - Sydney Children's Hospital Network - Randwick, Randwick, New South Wales
  - The Alfred, Melbourne, Victoria
- Canada (2):
  - Sunny brook Health Sciences Centre- Bayview Campus, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- France (7):
  - Institut Bergonie, Bordeaux, Aquitaine
  - Hôpital Nord de Marseille, Marseille, Bouches-du-Rhône
  - Hôpital Morvan, Brest, Finistère
  - Institut de Cancerologie de l'Ouest- Angers, Angers, Pays de la Loire Region
  - Gustave Roussy, Villejuif, Val-de-Marne
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse
  - Hôpital Universitaire Pitié Salpêtrière, Paris, Île-de-France Region
- Germany (3):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Krankenhaus Nordwest, Frankfurt am Main, Hesse
  - Charité - Universitätsmedizin Berlin, Berlin
- Italy (4):
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST, Meldola, Forli-Cesena
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli, Naples
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
- Norway (2):
  - Haukeland Univeritetssjukehus, Bergen, Hordaland
  - Oslo Universitetssykehus-Radiumhospitalet, Oslo
- South Korea (6):
  - Catholic University of Korea Saint Vincent's Hospital, Suwon, Gyeonggi-do
  - Seoul National University Hospital, Suwon, Gyeonggido
  - Dong-A University Hospital, Pusan, Gyeongsangnam-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Seoul National University Hospital, Seoul, Seoul Teugbyeoisi
  - Severance Hospital, Seoul, Seoul Teugbyeolsi
- Spain (6):
  - Hospital Clinico Universitarlo de Santiago, Santiago de Compostela, A Coruña
  - Hospital Clinico Universitarlo de Valencia, Valencia, Valencia
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Sweden (2):
  - Skånes Universitetssjukhus, Lund, Skåne County
  - Karolinska Universitetssjukhuset, Solna, Stockholm County
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester, England
  - Sarah Cannon Research Institute, London

IPD SHARING:
Plan to Share IPD: Yes
Fore is committed to sharing with qualified external researchers access to deidentified patient-level data and related study documents (eg. study protocol) from eligible studies following publication of the study results.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication of summary data and ending 36 months following article publication.
Access Criteria: Qualified external researchers may submit a request to access deidentified patient-level data and related study documents (eg. study protocol). These requests will be reviewed and approved by an independent committee on the basis of scientific merit and may be subject to certain criteria, conditions, and exceptions. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.